CLINICAL TRIAL: NCT02400385
Title: A Phase II Trial of Sunitinib and Nivolumab for KIT-mutated Advanced Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: With recent advances in immunotherapy scientific question not significant
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 703131-1
Record Dates: First submitted 2015-03-16; First posted 2015-03-27 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Sunitinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Sunitinib 50mg/day, 4 weeks on and 2 weeks off, and concurrent nivolumab 3mg/kg iv every 2 weeks, both for three years if tolerated.
  Interventions: Drug: sunitinib; Drug: nivolumab

INTERVENTIONS:
Drug: sunitinib — sunitinib 50mg/day po, 4 weeks on 2 weeks off
  Other Names: Sutent
Drug: nivolumab — nivolumab 3mg/kg IV ever 2 weeks
  Other Names: Opdivo

SUMMARY:
This will be a phase II trial of the combination of sunitinib and nivolumab in patients with advanced, measurable, metastatic melanoma who harbor mutations in the KIT gene in their tumors. It is a multi-center trial using the FDA-approved doses of both sunitinib and nivolumab. Sunitinib will be provided by Pfizer. Endpoint is RECIST response rate and PFS.

DETAILED DESCRIPTION:
Curtin and Bastian in 2006 first described KIT mutations in melanoma. Although uncommon in non-acral cutaneous melanoma, these mutations are frequent in mucosal and acral melanomas. The KIT mutations in melanoma are similar to the KIT mutations in gastrointestinal intestinal stromal sarcomas (GIST) and these are believed to be driver mutations. In melanomas these mutations occur in an exclusive pattern in tumors without NRAS, BRAF, or GNAQ mutations. There is evidence that stage four melanoma patients with KIT mutations have a worse prognosis than other patients with similar stage and primary site.

Both imatinib and sunitinib are FDA approved for treatment of patients with GIST; these and other oral tyrosine kinase KIT inhibitors have been studied in melanoma patients with KIT mutations. Imatinib is the best studied with objective responses in 20% of patients in a multicenter trial, considerably lower than the efficacy seen in GIST. Sunitinib has the theoretical advantage of anti-angiogenic activity as well as anti -KIT activity and demonstrated objective responses in three of four patients in a small trial sponsored by Pfizer.(see citation).

Immunotherapy has a major role in the treatment of metastatic melanoma, with the approval and use of both Interleukin-2 and ipilimumab because of the ability of immunotherapy to produce durable responses and prolonged survival in a minority, but a significant number, of patients . Both sunitinib and ipilimumab have intestinal perforation as an unusual but very significant toxicity, which argues against using those two agents in combination. The anti-PD-1 antibody Nivolumab, however, is an immunologic agent that yields rapid and durable responses in melanoma with less colitis and less risk of intestinal perforation than ipilimumab. Nivolumab was FDA approved in December 2014 and NCCN guidelines include it as a first-line option.

Combining KIT receptor inhibition with sunitinib with immunotherapy with Nivolumab is an attractive investigational approach as the combination should produce complementary and perhaps synergistic efficacy.

Asim et al reported at ASCO in June 2014 a phase one study of sunitinib and nivolumab for the treatment of metastatic renal cell cancer. Sunitinib (50 mg/day x 4 week, off 2 weeks and nivolumab at 2mg/kg or 5mg/kg q 3 weeks was administered to 33 patients. No dose-limiting toxicities were seen but grade 3-4 AEs were seen in 24 of 33 patients. The most common AEs were elevated ALT (18%), hypertension (15%) and hyponatremia (15%). Objective responses sere seen in 52% (17/33) indicating an "encouraging activity and a manageable safety profile" in patients with renal cell cancer. The Nivolumab dose of 5mg/kg Q 3 weeks (1.67mg/kg/week) on that study is slightly above the usual dose of 3mg/kg Q 2 weeks (1.5mg/kg/week).

Study Design:

This is an open-label multi-center phase 2 study of sunitinib and Nivolumab in combination in patients with KIT mutated metastatic melanoma. Study to begin after FDA approval of nivolumab Total number of study subjects will be approximately 12-18 patients.

Objectives

Primary objective:

1. To describe the preliminary clinical efficacy of sunitinib when given in combination with nivolumab to patients with KIT-mutated melanoma
2. To describe the immunologic effects of sunitinib when administered in combination with Nivolumab

Co-primary endpoints:

1. Objective response using RECIST 1.1 immune modified response criteria
2. Progression-free survival using immune-modified response criteria

Secondary endpoints:

1. Toxicities using CTAE criteria
2. Changes in peripheral blood total lymphocyte counts and T and B cell count
3. Overall survival The trial is sponsored by the California Pacific Medical Center Research Institute and the sunitinib will be provided by Pfizer. Commercial sources will be used for the nivolumab, whose use is in accord with NCCN guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable stage 3 or stage 4 metastatic melanoma
2. A mutation, translocation, or fusion in the KIT gene in the patient's tumor felt to be potentially sensitive to tyrosine kinase inhibition. Expression of CD113 or other immunohistochemical test will not by itself satisfy this requirement.
3. Evidence of measurable disease by RECIST criteria 1.2 Bone lesions, ascites, peritoneal carcinomatosis or miliary lesions, pleural or pericardial effusions, lymphangitis of the skin or lung, cystic lesions, or irradiated lesions are not considered measurable. .
4. Resolution of all acute toxic effects of prior radiotherapy or surgical procedures to NCI CTCAE Version 3.0 grade ≤1.
5. Adequate organ function as defined by the following criteria:

   * Absolute neutrophil count (ANC) ≥1,000/µL
   * Platelets ≥75,000/µL
   * Hemoglobin ≥8.0 g/dL
   * Serum calcium ≤12.0 mg/dL
   * Serum creatinine ≤1.5 x ULN
   * Total serum bilirubin ≤1.5 x ULN
   * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤2.5 x local laboratory upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to underlying malignancy
6. Karnofsky performance status > 60 %.
7. Male or female, 18 years of age or older.
8. Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to undergoing study screening procedures.
9. Subject's willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Brain metastasis requiring daily corticosteroid dosage over 7 .5mg/ day prednisone or equivalent.
2. Prior therapy with sunitinib or anti-PD-1 or anti-PDL-1 antibodies (pembrolizumab, nivolumab, etc.) Prior therapy with other KIT inhibitors (dasatinib, nilotinib, imatinib, etc.) allowed but results from these patients will be analyzed separately.
3. Major surgery or radiation therapy within 2 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
4. NCI CTCAE Version 3.0 grade 3 hemorrhage within 4 weeks of starting the study treatment.
5. Any of the following within the 4 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic heart failure, or cerebrovascular accident.
6. Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade > 2.
7. Prolonged QTc interval on baseline EKG (>450 msec for males or >470 msec for females)
8. Uncontrolled hypertension (> 170/100 mm hg despite optimal medical therapy).
9. Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g., QOL, are allowed.
10. Concomitant treatment with a drug having proarrhythmic potential (terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide and flecainide)
11. Use of potent CYP3A4 inhibitors and inducers 7 and 12 days before dosing, respectively (see below).
12. Definite history of ulcerative colitis or Crohn's disease or lupus
13. History of allogeneic transplant.
14. Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Objective response by RECIST 1.1 | 3 years

SECONDARY OUTCOMES:
Grade 3, 4, or 5 adverse events in patients on trial | 3 years
  Adverse events will be measured and recorded using CTAE criteria.
Change in peripheral blood lymphocytes | 3 years
  Change in total and lymphocyte subsets in select patients
Progression-free survival by RECIST | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David R Minor, M.D., Study Chair — California Pacific Medical Center Research Institute; Kevin B Kim, MD, Principal Investigator — California Pacific Melanoma Center
Locations (1):
- California Pacific Medical Center Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minor DR, Kashani-Sabet M, Garrido M, O'Day SJ, Hamid O, Bastian BC. Sunitinib therapy for melanoma patients with KIT mutations. Clin Cancer Res. 2012 Mar 1;18(5):1457-63. doi: 10.1158/1078-0432.CCR-11-1987. Epub 2012 Jan 18. PMID 22261812